CLINICAL TRIAL: NCT05614726
Title: Effects of a Probiotic Supplement on Gastrointestinal Symptoms and Microbiome Modulation
Brief Title: A Probiotic Blend Reduces Gastrointestinal Symptoms and Positively Impacts Microbiota Modulation in a Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Applied Health Sciences, LLC (Industry)
Collaborators: Biohm Health, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-CAHS-102
Record Dates: First submitted 2022-11-05; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Microbiota; Constipation; Candida
MeSH Terms: conditions — Constipation; Torulopsis | interventions — Lacteol; alpha-Amylases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Consists of 575 mg rice oligodextrin
  Interventions: Dietary Supplement: 575mg [30 billion colony forming units] probiotic blend of Bifidobacterium breve, Lactobacillus acidophilus, Lacticaseibacillus rhamnosus, Saccharomyces boulardii, and alpha amylase
- Active (Active Comparator): Consists of 575mg [30 billion colony forming units probiotic blend of Bifidobacterium breve 19bx, Lactobacillus acidophilus 16axg, Lacticaseibacillus rhamnosus 18fx, Saccharomyces boulardii 16mxg, and alpha amylase
  Interventions: Dietary Supplement: 575mg [30 billion colony forming units] probiotic blend of Bifidobacterium breve, Lactobacillus acidophilus, Lacticaseibacillus rhamnosus, Saccharomyces boulardii, and alpha amylase

INTERVENTIONS:
Dietary Supplement: 575mg [30 billion colony forming units] probiotic blend of Bifidobacterium breve, Lactobacillus acidophilus, Lacticaseibacillus rhamnosus, Saccharomyces boulardii, and alpha amylase — A multi-strain probiotic blend

SUMMARY:
This randomized, placebo-controlled, double-blind study will determine the effect of daily supplementation with a probiotic blend in 60 apparently healthy men and women recruited at a single investigational center in Northeast Ohio (i.e., The Center for Applied Health Sciences).

Subjects will attend three study visits. During Visit 1, subjects will be screened for participation [i.e., medical history, routine blood work, background baseline diet]. During Visits 2 and 3 subjects will complete questionnaires that assess their gastrointestinal health (e.g., abdominal discomfort/bloating, constipation, regularity, stool consistency). Visits 2 and 3 will correspond to before (week 0) and after six weeks of supplementation, respectively, with the probiotic dietary supplement or placebo.

ELIGIBILITY:
Inclusion Criteria:

* all participants were required to be between 30-60yr
* score ≥12 on the GSRS
* have a body mass ≥120 pounds (54.5kg)
* body mass index (BMI) between 20.0-34.99kg/m2
* normotensive (<140/<90mmHg)
* normal resting heart rate (<90bpm)

Exclusion Criteria:

* Female participants who were pregnant or nursing
* history of unstable or new-onset cardiovascular or cardiorespiratory disease;
* stroke, diabetes, or other endocrine disorder;
* use of any nutritional supplement known to alter the gut microbiota/microflora;
* use of probiotic supplements or prebiotic supplements in the previous 4 weeks and for the duration of the study;
* use of any antibiotics, antifungals, antivirals, or antiparasitic within 8 weeks of the start of the study or throughout the study;
* any changes in diet within 4 weeks of study start date or throughout study duration;
* if the participant was unwilling to abstain from gut altering supplements for the study;
* malignancy in the previous 5yr except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin);
* prior gastrointestinal bypass surgery (i.e., Lapband);
* any known gastrointestinal or metabolic diseases that might impact nutrient absorption or metabolism [e.g. short bowel syndrome, diarrheal illnesses, history of colon resection, gastroparesis, Inborn-Errors-of-Metabolism (such as PKU)];
* any chronic inflammatory condition/disease (e.g. rheumatoid arthritis, Crohn's disease, ulcerative colitis, Lupus, HIV/AIDS, etc.);
* known sensitivity to any ingredient in the test formulations as listed in the certificates of analysis.
* currently participating in another research study with an investigational product or had participated in another research study in the past 30 days
* any other diseases/conditions that, in the opinion of the medical staff, could confound the primary endpoints or place the subject at increased risk of harm if they were to participate.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Flatulence (gas) | Change from baseline to 6 weeks.
  Flatulence (gas) as measured by a 10 cm visual analogue scale, where higher values represent greater flatulence.
Gastro-intestinal bloating | Change from baseline to 6 weeks.
  Gastro-intestinal bloating as measured by a 10 cm visual analogue scale, where higher values represent greater bloating.
Abdominal discomfort | Change from baseline to 6 weeks.
  Abdominal discomfort as measured by a 10 cm visual analogue scale, where higher values represent greater discomfort.
Gastrointestinal Symptom Rating Scale (GSRS) | Change from baseline to 6 weeks.
  Gastrointestinal problems as measured by the GSRS questionnaire, where higher values represent increased severity of gastrointestinal problems.

SECONDARY OUTCOMES:
Stool consistency | Change from baseline to 6 weeks.
  Stool consistency as measured by a 10 cm visual analogue scale, where higher values represent harder stools.
Stool regularity | Change from baseline to 6 weeks.
  Stool regularity as measured by a 10 cm visual analogue scale, where higher values represent more regular stools.
Constipation | Change from baseline to 6 weeks.
  Constipation as measured by a 10 cm visual analogue scale, where higher values represent more greater constipation.

OTHER OUTCOMES:
Short Form Health Survey (SF-36) | Change from baseline to 6 weeks.
  Health status as measured with the SF-36 questionnaire, where scores range from 0 to 100, and higher values represent better health status.

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Applied Health Sciences, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] La Monica MB, Raub B, Lopez HL, Ziegenfuss TN. A probiotic amylase blend reduces gastrointestinal symptoms in a randomised clinical study. Benef Microbes. 2023 Oct 23;14(5):459-476. doi: 10.1163/18762891-20230043. PMID 38350481